CLINICAL TRIAL: NCT03624335
Title: Influence of Umbilical Cord Clamping Time in the Newborn, Secondary Neonatal Morbidity and Iron Deposits in the Neonate
Brief Title: Influence of Umbilical Cord Clamping Time in the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pascual Gregori Roig (Other)
Collaborators: Hospital Universitario de la Plana (Other); FUNDACIÓN DAVALOS FLETCHER (Unknown)
Responsible Party: Sponsor-Investigator, Pascual Gregori Roig, Adjunct Pediatrician of University Hospital of La Plana (Spain), Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CORD STUDY
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Anemia Neonatal; Polycythemia Secondary; Hyperbilirubinemia, Neonatal
Keywords: Umbilical cord clamping; Anemia Neonatal; Iron metabolism disorders
MeSH Terms: conditions — Anemia, Neonatal; Hyperbilirubinemia, Neonatal; Iron Metabolism Disorders | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Randomised controlled trials comparing early and late cord clamping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: ECC (Experimental): In the ECC group, the cord was clamped immediately after delivery, before the first minute of life.
  Blood test 6hours after clamping Blood test 24hours after clamping Blood test 48hours after clamping Blood test 28days after clamping
  Interventions: Procedure: ECC; Procedure: Blood Test 6hours; Procedure: Blood Test 24hours; Procedure: Blood Test 48hours; Procedure: Blood Test 28days
- Group 2: DCC (Experimental): In the DCC group, the cord was clamped when it stops beating. Blood test 6hours after clamping Blood test 24hours after clamping Blood test 48hours after clamping Blood test 28days after clamping
  Interventions: Procedure: DCC; Procedure: Blood Test 6hours; Procedure: Blood Test 24hours; Procedure: Blood Test 48hours; Procedure: Blood Test 28days

INTERVENTIONS:
Procedure: ECC — Early clamping of the umbilical cord
  Arms: Group 1: ECC
Procedure: DCC — Delayed clamping of the umbilical cord
  Arms: Group 2: DCC
Procedure: Blood Test 6hours — Blood Test 6hours
Procedure: Blood Test 24hours — Blood Test 24hours
Procedure: Blood Test 48hours — Blood Test 48hours
Procedure: Blood Test 28days — Blood Test 28days

SUMMARY:
This study compares two umbilical cord clamping times; the early one, up to a minute (ECC) and the late or delayed one, when the cord stop beating (DCC). The additional blood volume delivered to the newborn from the placenta - placental transference - by delaying umbilical cord ligation, increases the contribution of neonatal iron with increased iron stores in the infant, without increasing neonatal morbidity.

DETAILED DESCRIPTION:
It is an intervention study without drugs administration with a longitudinal, prospective comparison and correlational design.

Patients are recruited by simple random sampling to one of the two intervention groups:

Group 1-ECC: Early clamping of the umbilical cord (before the first minute of life).

Group 2-DCC: Delayed clamping of the umbilical cord (when it stops beating).

ELIGIBILITY:
Inclusion Criteria:

- neonates with a gestational age of 35 to 42 weeks and born through normal vaginal delivery.

Exclusion Criteria:

* monochorionic multiples
* incarcerated mothers
* placenta previa
* concern for abruptions
* Rh sensitization
* hydrops
* congenital anomalies
* the obstetrician declining to perform the intervention

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
haemoglobin | 6hours
  haemoglobin level
haemoglobin | 28 days
  haemoglobin level
haematocrit | 6 hours
  haematocrit level
haematocrit | 28 days
  haematocrit level

SECONDARY OUTCOMES:
serum ferritin | 6hours
  serum ferritin level
serum ferritin | 28days
  serum ferritin level
bilirubin | 6hours
  bilirubin level
bilirubin | 28days
  bilirubin level

CONTACTS AND LOCATIONS:
Overall Officials: Vanesa Rodenas, PhD, Study Chair — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Hospital Universitario de La Plana, Villarreal, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Protocol study & Data Analysis

REFERENCES:
- [Derived] Orenga-Orenga BJ, Gregori-Roig P, Real-Fernandez A, Donat-Colomer F, Sanchez-Thevenet P. Umbilical cord clamping time and maternal satisfaction. Midwifery. 2022 Dec;115:103487. doi: 10.1016/j.midw.2022.103487. Epub 2022 Sep 13. PMID 36126369